CLINICAL TRIAL: NCT06374498
Title: Study to Determine the Clinical Significance of Intravascular OCT-NIRAF
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Guillermo Tearney, Professor of Pathology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023P003247
Record Dates: First submitted 2024-03-25; First posted 2024-04-18 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Cardiovascular Diseases; Coronary Artery Disease
Keywords: Optical Coherence Tomography; NIRAF; Cardiovascular; CAD
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Participants with stable CAD or acute coronary syndromes undergoing invasive coronary angiography (Experimental): Participants referred to the Cardiology Division of the Massachusetts General Hospital, undergoing coronary angiography for stable or acute coronary disease and eligible for percutaneous coronary intervention (PCI) will be eligible for the study.
  Interventions: Device: OCT-NIRAF

INTERVENTIONS:
Device: OCT-NIRAF — Subjects will be imaged with OCT-NIRAF research catheter during their clinically indicated coronary angiogram. In addition, the subject will also receive two Coronary Computed Tomography Angiography (CCTA) 12 months apart, and images will be analyzed.

SUMMARY:
Participants undergoing coronary angiography for stable or acute coronary disease presentations and eligible for percutaneous coronary intervention (PCI) will be imaged with OCT-NIRAF at baseline and with CCTA 12 months apart to demonstrate that:

1. NIRAF coronary artery signal level (patient, artery, lesion basis) is correlated with the severity of coronary artery disease.
2. NIRAF coronary artery signal level is a predictor of plaque progression on a per participant, per artery, or per lesion basis.

DETAILED DESCRIPTION:
This study will provide preliminary data on the clinical value of intracoronary OCT-NIRAF imaging in participants undergoing invasive coronary angiography in the cardiac catheterization laboratory. This is a single site, prospective feasibility study where 40 study subjects undergoing coronary angiography for stable or acute coronary disease presentations and eligible for percutaneous coronary intervention (PCI) will undergo intravascular imaging, including standard-of-care IVUS and then OCT-NIRAF pullback imaging conducted during an iodinated contrast flush. Patients will be consented prior to catheterization. Participant characteristics such as age, sex, BMI, and current medication regimen will be recorded. Standard of care blood chemistry will be reviewed and lab values from the subject's electronic medical records will be input into the study's Case Report Form when available. A complete medical history and data regarding prescribed cardiac medications also be transcribed from the EMR into the CRF.

Coronary Angiography will be performed. For participants for whom coronary angiography provides a clinical indication for intravascular imaging or PCI without any exclusion criteria, 40 study participants will undergo intravascular imaging, including standard-of-care IVUS and then research study OCT-NIRAF pullback imaging, conducted during an iodinated contrast flush.

Intravascular imaging of the PCI target artery will be done prior to PCI unless the interventional cardiologist determines that intervention is required to deliver the imaging catheters. The other major coronary arteries may also be imaged by IVUS and OCT-NIRAF based on clinical assessment of the appropriateness of imaging by the interventional cardiologist.

In addition, participants will obtain a baseline coronary CTA at MGH, using standard clinical protocols in the MGH Department of Radiology.

Follow up imaging: After 12 months (+/- 28 days), participants will undergo a follow-up study coronary CTA, to assess for plaque progression compared to the baseline coronary CTA.

Follow up: Participants will undergo standard-of-care cardiology follow-up and medical record review follow-up by study staff at 1 month (+/- 7 days), 6 months (+/- 28 days), and 1 year (+/- 28 days). After completion of the CCTA and final telephone 12-month follow-up, patients will be released from the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with stable CAD or acute coronary syndromes undergoing invasive coronary angiography in the MGH cardiac catheterization laboratory
* Participant is eligible for PCI
* Participants must be over the age of 18
* Participant must be able to give informed consent
* Women with childbearing potential must have a negative pregnancy test within seven days prior to the procedure

Exclusion Criteria:

* CLINICAL EXCLUSION CRITERIA:

  * Renal insufficiency (GRF<45 ml/min/1.73m2)
  * Pregnancy
  * Acute myocardial infarction: Participants with ST elevation MI will be excluded for at least 72 hours post event. Participants with non-ST elevation MI will be excluded if they have evidence of ongoing ischemia defined as chest pain or new ECG changes in the previous 12 hours and/or rising cardiac biomarker enzymes (e.g., troponin or CKMB)
  * Evidence of ongoing or active clinical instability, including acute chest pain (sudden onset), cardiogenic shock, unstable blood pressure with systolic blood pressure <90 mmHg, and severe congestive heart failure (NYHA III or IV) or acute pulmonary edema,
  * Emergent procedures
  * Ejection fraction <= 35%
  * Clinically significant bleeding within the past 14 days
  * Any active, serious, life-threatening disease with a life expectancy of less than 12 months
  * Inability to be evaluated at follow-up
  * Currently enrolled in another study utilizing OCT imaging, or in an investigational trial that involves a non-approved cardiac drug or device
  * Participants under the protection of justice, guardianship, or curatorship

CARDIAC CATHETERIZATION LABORATORY - EXCLUSION CRITERIA (AFTER DIAGNOSTIC CORONARY ANGIOGRAM):

* Participant deemed not indicated for intravascular imaging or PCI
* Inability to perform intravascular imaging of a target artery
* Left main disease >= 50% stenosis in participants that do not have a functioning LAD bypass graft
* Clinical instability that develops after IVUS imaging but prior to OCT-NIRAF imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Plaque size estimation using OCT-NIRAF | Data will be analyzed within 1 year after the procedure.
  Optically derived signatures (OCT-NIRAF) will be compared to plaque volume measured by CCTA at baseline.
Plaque progression estimate using OCT-NIRAF | Data will be analyzed within 1 year after the procedure.
  Changes in plaque volume will be measured by CCTA at baseline and after 1 year. Optically derived signatures (OCT-NIRAF) obtained at baseline will be compared to changes in plaque volume.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo J Tearney, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No